CLINICAL TRIAL: NCT02636569
Title: Topical Chemoprevention of Skin Cancer Biomarkers
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: National Cancer Institute (NCI) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Principal Investigator, Craig Elmets, Immediate Past Chairman and Professor Emeritus of Dermatology, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: F150814005; 2015678 (Other Grant/Funding Number: National Health Institute)
Record Dates: First submitted 2015-12-17; First posted 2015-12-22 (Estimated); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Non-melanoma Skin Cancer
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- diclofenac once daily (Active Comparator): Topical diclofenac, will will be applied onto the skin of one arm, every day for 30 days. Enough medication will be used to cover an area of approximately 4 square inches( a 2 inch by 2 inch square). The medications will come in a tube. The medications will be applied to the same sun exposed site on the arm every day. The research team will provide instructions for the correct application of the treatment.
  Interventions: Drug: topical diclofenac daily
- placebo (Placebo Comparator): The topical medication will will be applied onto the skin of one arm, once daily for 30 days. Enough placebo will be used to cover an area of approximately 4 square inches( a 2 inch by 2 inch square). The placebo will come in a tube. The placebo will be applied to the same sun exposed site on the arm every day. The research team will provide instructions for the correct application of the treatment.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: topical diclofenac daily — Topical diclofenac will be applied daily for 30 days. Each subject will be seen for a screening visit as well as a baseline visit and a visit at month 1. As part of the study small biopsies will be taken from three locations at the baseline visit. The biopsy will be taken from one actinic keratosis, one sun exposed area and one not sun exposed area. A biopsy is a small surgical procedure where a small piece of your skin is removed.
  After applying the medications for 30 days you will return to the clinic for your 30 day visit. At this visit you will again have three biopsies taken; one AK, one sun exposed, and one non sun exposed.
  Other Names: topical diclofenac
  Arms: diclofenac once daily
Drug: placebo — placebo Each subject will be seen for a screening visit as well as a baseline visit and a visit at month 1. As part of the study small biopsies will be taken from three locations at the baseline visit. The biopsy will be taken from, one actinic keratosis, one area that is typically exposed to the sun as well as a site that is typically protected from sun light. A biopsy is a small surgical procedure where a small piece of your skin is removed.
  After applying the medications for 30 days you will return to the clinic for your 30 day visit. At this visit you will again have two biopsies taken. One of these biopsies will be from the skin on your arm that was treated with medication for the prior 30 days, and the other biopsy will be from a site that typically is not exposed to the sun.
  Arms: placebo

SUMMARY:
This research study will test how well one topical medications work to prevent the development of non-melanoma skin cancers by reversing certain biomarkers in the skin. This study is also looking at the optimal dose of a medication in a small number of people. Biomarkers are molecules that are found in the body and inside of cells. Some biomarkers are associated with specific diseases such as skin cancer. In this study, one topical medication will be evaluated; diclofenac. Diclofenac and is approved by the Food and Drug Administration (FDA) for other uses. 24 patients will be enrolled in this study by University of Alabama at Birmingham.

DETAILED DESCRIPTION:
Men and women (≥ 18 yo)who have been seen as patients in the Dermatology Clinic at the University of Alabama at Birmingham with a history of basal cell or squamous cell carcinoma of the skin and at least 8 actinic keratoses on the upper extremities are potentially eligible for study participation.

We propose to examine one topical medication which is already FDA approved,with a placebo comparator. The purpose of the study is to see if diclofenac applied daily will affect levels of specific biomarkers in the skin that are associated with risk of developing skin cancer. We hope to see these levels decrease with once daily use of this medication. Results from this study will help guide us in a second study where we will look at longer term use of these medications and how they are associated with changes in skin biomarkers that are related to skin cancer. The second longer study will use the dose (once or twice daily topical application of diclofenac and DMFO) that resulted in a decrease in biomarkers, as discovered in this currently proposed study.

ELIGIBILITY:
Inclusion Criteria:

o Ability to understand and willingness to sign a written informed consent document

* ECOG performance status 0-1
* Willing and able to participate for the full duration of the study
* Greater than 4 weeks from:

Prior major surgery for any indication Prior chemotherapy, hormonal therapy or radiation therapy for cancer o Willing to abstain from: The application of topical medications including prescription and over the counter preparations (e.g. Topical preparations containing corticosteroids or vitamin A derivatives) to areas of actinic damage for the duration of the study. Use of moisturizers/emollients and sunscreens on these areas is allowed.

Chronic (defined as > 3 times/week for more than 2 consecutive weeks/year) NSAID and COX-2 inhibitor use (other than cardioprotective doses of aspirin < 100 mg po QD) for the duration of the study. For routine analgesia, subjects may take acetaminophen as necessary.

* Normal organ and marrow function defined as laboratory values falling within the specified ranges for the following tests (performed within 14 days of registration) Hematologic • WBC > 3,000/ul • Hemoglobin > lower limit of normal • Platelet count > 100,000/ul Hepatic

  • Total bilirubin < 1.5 X ULN

  • AST (SGOT) < 1.5 X ULN
  * ALT (SPGT) < 1.5 X ULN Renal
  * Serum creatinine < 1.5 X ULN
  * BUN < 1.5 X ULN
* Females of childbearing potential must:

Have been using adequate contraception (abstinence, IUD, birth control pills or spermicidal gel with diaphragm or condom) since their last menses Have a documented negative serum pregnancy test within 14 days prior to the first dose of study medication Females are not considered to be of childbearing potential if they are at least 1 year post-menopausal or have had a tubal ligation, bilateral oophorectomy or hysterectomy.

o The effects of topical DFMO + topical diclofenac on the developing fetus are unknown. Therefore all females of childbearing potential must agree to use adequate contraception (abstinence, IUD, birth control pills, or spermicidal gel with diaphragm or condom) for the duration of study participation.

Exclusion Criteria:

o Within 6 months prior to randomization: Use of oral or intravenous corticosteroids for more than 2 consecutive weeks Use of inhaled corticosteroids for more than 4 consecutive weeks

o Any of the following in the 4 weeks (or as indicated) prior to randomization: Major surgery for any indication Cytotoxic chemotherapy for any indication (including methotrexate for arthritis) Anti-cancer treatment of any type other than for a stage 0-2 non-melanoma skin cancer Hormonal therapy for cancer prevention (including tamoxifen) Note: treatment with finasteride/dutasteride for BPH does not render a participant ineligible.

Radiation therapy Topical medications for the treatment of actinic keratosis or skin cancer (retin A, 5-FU, imiquimod) in the 6 months prior to randomization.

Laser resurfacing, dermabrasion, cryotherapy, chemical peel and electrodissection ± curettage in the 6 months prior to randomization.

Nasally inhaled corticosteroids (except mometasone - Nasonex) Aspirin (>100 mg/day) - Note: cardioprotective doses (< 100mg/day) are acceptable.

NSAIDs (other than aspirin < 100mg/day) or COX-2 inhibitors > 3 times/week for more than a two week period Topical steroids

o Any personal history of: Invasive cancer diagnosed or treated within the past 5 years. Participants who have been in remission for 5 years or more and have not required treatment in the past 5 years may be eligible if the principal investigator believes there is little to no risk of recurrence.

Solid organ or bone marrow transplant Keloid formation Photosensitivity disorder Hypersensitivity or adverse reactions to nonsteroidal anti-inflammatory agents or to DFMO Any disease that predisposes to NMSC An immunodeficiency disorder or the use of an immunosuppressive drug Any skin disease that would interfere with interpretation of results

* Any family history of Ornithine diaminotransferase deficiency in a first degree relative
* Concurrent use of the following medications or treatments Anticoagulants including warfarin and heparin Other NSAIDs (other than aspirin <100 mg/day) on a daily basis Topical chemotherapy, cryotherapy, radiotherapy or any other skin lesion treatment to areas of skin being followed in this study Systemic therapy with psoralens, immunotherapy, retinoids, or radiation therapy Cytotoxic chemotherapy for any reason (including methotrexate for arthritis) Laser resurfacing, dermabrasion or chemical peels Topical or systemic immunosuppressive therapy.
* Females who are pregnant or lactating. Should a woman become pregnant or suspect she is pregnant while she is participating in this study she should notify the study physician immediately.
* Uncontrolled concurrent illness including ongoing or active infection, psychiatric illness/social situations that would limit compliance with study requirements or other underlying serious medical condition which, in the investigator's opinion, might preclude study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2017-10-25 (Actual); Primary Completion 2025-12-01 (Actual); Study Completion 2025-12-31 (Actual)

PRIMARY OUTCOMES:
Optimal Dosing of topical diclofenac and topical DFMO for the reduction of non melanoma skin cancer biomarkers | 1 year
  The primary outcome measure will be to determine whether subjects randomized to topical diclofenac ± topical DFMO will have a significant reduction (≥40% reduction, p ≤ 0.05) in skin biomarkers associated with development of non melanoma skin cancers after treatment once daily, twice daily or with placebo.
Optimal Dosing of topical diclofenac and topical DFMO for the reduction of actinic keratoses | 1 year
  A secondary outcome will be to determine whether subjects randomized to diclofenac ± DFMO will have fewer actinic keratoses at the end of treatment once daily, twice daily or with placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Craig Elmets, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham Whitaker Clinic, Birmingham, Alabama, United States